CLINICAL TRIAL: NCT07055178
Title: A Perioperative Virtual Reality Intervention for Pain and Anxiety Management During Vasectomies: A Randomized Controlled Trial
Brief Title: Perioperative Virtual Reality Intervention for Pain and Anxiety During Vasectomies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Renée El-Gabalawy, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS26972
Record Dates: First submitted 2025-06-13; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Vasectomy; Pain; Anxiety; Virtual Reality
Keywords: Virtual Reality; TRIPP; Vasectomy
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Vasectomy (Active Comparator): Vasectomy treatment as usual, with local anesthetic, without virtual reality.
  Interventions: Other: Treatment as usual
- Virtual Reality Vasectomy (Experimental): This group of participants will receive undergo their vasectomy with the virtual reality intervention alongside the local anesthetic.
  Interventions: Device: Virtual reality (VR) guided meditation therapy

INTERVENTIONS:
Device: Virtual reality (VR) guided meditation therapy — Participants will engage in the TRIPP relaxation app on the MetaQuest 3 VR headset.
  Arms: Virtual Reality Vasectomy
Other: Treatment as usual — Participants undergo a standard vasectomy.
  Arms: Standard Vasectomy

SUMMARY:
The goal of this clinical trial is to learn if a virtual reality (VR) program (TRIPP) can reduce pain, anxiety, and distress in adult men (aged 18+) undergoing a vasectomy under local anesthesia. The main questions it aims to answer are:

* Does using VR during a vasectomy lower patients' pain during the procedure compared to standard care?
* Does VR reduce anxiety and distress compared to standard care?
* Are patients more satisfied with their experience when using VR compared to standard care?

Researchers will compare two groups:

* VR group: Patients will use a VR headset with a guided meditation program (TRIPP) during their vasectomy.
* Control group: Patients will receive standard care (no VR).

Participants will:

* Be randomly assigned to either the VR group or control group.
* Complete brief questionnaires before, during, and after the procedure (about 15-20 minutes each time).
* (VR group only) Use a VR headset during the procedure and provide optional feedback about the experience.

Why is this important? Vasectomies are typically done with local anesthesia (pain relief), but many patients still feel anxiety or discomfort. VR may help distract and relax patients, improving their experience. This study will help health professionals understand if VR could be a useful option for future patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Can speak and read English.
* Have elected for a vasectomy.
* Are scheduled to undergo their vasectomy under local anesthesia at the Men's Health Clinic

Exclusion Criteria:

* Those who are not competent to provide informed consent (e.g., due to cognitive impairment).
* Those who are unable to participate in a VR intervention (e.g., due to visual or auditory impairment).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) for Pain Severity | Perioperatively (midway through procedure) and immediately following the procedure.
  During and immediately following the procedure, patients will be momentarily interrupted to give a brief NRS verbal response question measure of their level of acute pain, this is on a scale of 0-10; 10 = most severe pain.

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) for Discomfort Severity | Perioperatively (midway through procedure) and immediately following the procedure.
  During and immediately following the procedure, patients will be momentarily interrupted to give a brief NRS verbal response question measure of their level of acute discomfort, this is on a scale of 0-10; 10 = most severe pain.
Numeric Rating Scale (NRS) for Anxiety Severity | Perioperatively (midway through procedure) and immediately following the procedure.
  During and immediately following the procedure, patients will be momentarily interrupted to give a brief NRS verbal response question measure of their level of acute anxiety, this is on a scale of 0-10; 10 = most severe pain.
PROMIS Pain Intensity Scale Total Score | Within 10 minutes postoperatively (in the recovery room)
  Immediately following the procedure, patients will be asked to respond to a short verbal Patient-Reported Outcomes Measurement Information System (PROMIS) pain intensity questionnaire with questions surrounding experienced pain (scored 3 - 15 ; 15 = greatest pain severity).
State Trait Anxiety Inventory Total Score | 10 minutes preoperatively (baseline) and within 10 minutes postoperatively (in the recovery room.
  Brief self-report questionnaire with questions surrounding anxiety traits (scale 0-63 ; 63 = most severe anxiety)
National Comprehensive Cancer Network (NCCN) Anxiety Thermometer Score (adapted from Distress Thermometer) | 10 minutes preoperatively (baseline) and within 10 minutes postoperatively (in the recovery room.
  Brief self-report visual analogue scale (VAS) for anxiety. Scored from 0-10 ; 10 = extreme anxiety.
Satisfaction with Surgery | Within 10 minutes postoperatively (in the recovery room).
  Brief self-report item to assess overall satisfaction with their procedure. Scaled from 0-10 ; 10 = greatest satisfaction.
iGroup Presence Questionnaire (IPQ) Score | Within 10 minutes postoperatively (in the recovery room).
  Brief self-report questionnaire with several questions surrounding VR experience (spatial presence, involvement, and experience realism). Each question is scored independently on a 7-point Likert scale (from -3 to +3).
Virtual Reality Impressions Scale | Within 10 minutes postoperatively (in the recovery room).
  Brief self-report questionnaire with several questions surrounding the virtual reality program experience (spatial presence, involvement, and experience realism). Each question is scored independently on a 0 - 10 scale ; 0 = complete disagreement, 10 = complete agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Renée El-Gabalawy, MA, PhD, C. Psych, Principal Investigator — University of Manitoba; Premal Patel, MD, FRCSC, Principal Investigator — Manitoba Men's Health Clinic; Ahmed M Zalam, B.Sc., Principal Investigator — University of Manitoba
Locations (1):
- Manitoba Men's Health Clinic, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
Study data and information from the study will not be sent outside of the University of Manitoba. Records containing health related information will be treated as confidential in accordance with Personal Health Information Act of Manitoba (PHIA). Information gathered in this research study may be published or presented in public forums, however names and other identifying personal information will not be revealed. Data will be coded and names will not be released.